CLINICAL TRIAL: NCT05403814
Title: Mixed Reality Prototype of Multimodal Screening for Early Detection of Cognitive Impairments in Elderly: Protocol Development and Usability Study
Brief Title: Test and Usability of Mixed-reality Screening Tool for Early Detection of Cognitive Declines
Acronym: SCOBES-AR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: FH Joanneum Gesellschaft mbH (Industry)
Responsible Party: Sponsor
Other Study IDs: SCOBES-AR Validation Study 2
Record Dates: First submitted 2022-05-05; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Aging; Cognitive Change
Keywords: mixed reality; multimodal screening; cognitive impairment; smart cognition
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational screening procedure (no intervention) — observational screening procedure (no intervention)

SUMMARY:
The aim of this study as part of the SCOBES-AR project is to establish and test a protocol for implementation and usability of mixed reality-enhanced multidisciplinary screening tool for early detection of cognitive impairments in the elderly.

DETAILED DESCRIPTION:
Early diagnosis of cognitive impairments is an important step in the adequate management of dementia. The project "Smart Cognition & Behavior Screening powered by Augmented Reality" (SCOBES-AR) aims to develop a multimodal screening tool (MST) for early detection of cognitive impairments using augmented and virtual reality. In the first project phase validated assessments were selected, combined in MST and tested in 174 healthy elderly adults. In the present project phase, the developed MST will be partly enhanced by mixed reality (MR). This MR-enhanced prototype of screening tool (MR-MST) will be tested and compared to the previously developed MST. In addition, the usability of this enhanced prototype will be examined.

The study aims to establish a protocol for implementation and usability of MR-enhanced multidisciplinary screening tool for early detection of cognitive impairments in the elderly.

In this cross-over design study protocol 100 healthy participants (aged 60-75years) will be screened for cognitive declines using: i) specially developed MST (assessment of cognitive functions, olfactory sensitivity, nutritional preferences, gait parameters, reaction times, activities of daily living, and ii) MR-enhanced MST in which the assessments of cognitive functions, reaction time, activities of daily living and gait are performed using tailor made software and augmented reality and virtual reality hardware. The results of the MR-enhanced MST will be compared with those without MR. The usability of the developed MR-enhanced MST will be tested on 10 investigators and 10 test participants using observed summative evaluation and the co-discovery method and on 2 usability experts using the co-discovery method.

This study was funded by the Austrian Research Promotion Agency and received Ethic Vote from the Ethic committee of the Medical University of Graz. The MR-MST prototype and the study protocol for the present study were developed. To date, no results are available for this study protocol.

The development of the MR-MST prototype enables identifying best practise procedure for evaluating cognitive declines in the elderly using multimodal and MR-enhanced model.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 60-75 years
* Interest in participating in the study
* Signed written informed consent form

Exclusion Criteria:

* Clinical diagnosis of mild cognitive impairment or dementia
* Clinical diagnosis of mental illness (e.g. depression, psychosis)
* Reduced mobility (walking aid, wheelchair)
* Aided hearing or visual impairment
* Participation in any other cognitive training study within the last 6 months
* Present guardianship according to the provisions of the Austrian adult protection law

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of the city of Graz and Graz suburbs
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Brief Smell Identification Test. | Day 1.
  The test evaluates the olfactory functions. Scale 0-12 points: higher values indicate better olfactory performance.
Food-Frequency-Index. | Day 1.
  This assessment evaluates the dietary behavior. Dietary behavior is classified as poor (< 32 points), moderate (32-34 points), good (35-39 points), and very good (> 39 points).
Dementia-Detection-Test. | Day 1.
  The test evaluates the cognitive functions (recall of word list, number transcoding, semantic word fluency, digit span reverse).
  Scale 0-18 points: probability of dementia (0-8 points), light cognitive changes (9-12 points), healthy (13-18 points).
Erlangen Test of Activities of Daily Living in Persons with Mild Dementia or Mild Cognitive Impairment: items "mobility" and "finances", performed with pen-and-paper. | Day 1.
  For each of the 2 items ("mobility" and "finances") a score 0-6 points is given. Higher score indicates better performance.
Erlangen Test of Activities of Daily Living in Persons with Mild Dementia or Mild Cognitive Impairment: items "mobility" and "finances", performed with Virtual Reality. | Day 1.
  For each of the 2 items ("mobility" and "finances") a score 0-6 points is given using tailor-made software. Higher score indicates better performance.
Trail-Making Test, performed with pen-and-paper. | Day 1.
  The test evaluates the cognitive abilities and consists of two parts: connecting numbers and connecting numbers and letters in ascending order. The time (sec.) to perform the task is measured using a stop watch. Shorter time indicates better performance.
Trail-Making Test, performed with Augmented Reality. | Day 1.
  The test evaluates the cognitive abilities and consists of two parts: connecting numbers and connecting numbers and letters in ascending order. The time (sec.) to perform the task is measured using a tailor-made software. Shorter time indicates better performance.
Reaction Time Test, performed with contact plates. | Day 1.
  The test evaluates the complex reactivity (eye-hand, eye-leg and eye-hand-leg reactions) in response to visual signals displayed in a randomized order. The time (sec.) to perform the task is measured using a stop watch. Shorter time indicates better performance.
Reaction Time Test, performed with smartphone mobile application. | Day 1.
  The test evaluates the complex reactivity (eye-hand, eye-leg and eye-hand-leg reactions) in response to visual signals displayed in a randomized order. The time (sec.) to perform the task is measured using mobile application. Shorter time indicates better performance.
Dual Task Assessments, performed with direct observation. | Day 1.
  The assessment measures the influence of a cognitive task on gait parameters. Time to complete the task (sec.), number of steps and walking speed (steps/min.) will be calculated for the single task (walking) and the double task (walking and counting). Bigger difference between the parameters in both tasks indicates cognitive declines.
Dual Task Assessments, performed with Augmented Reality. | Day 1.
  The assessment measures the influence of a cognitive task on gait parameters. Time to complete the task (sec.), number of steps and walking speed (steps/min.) will be calculated for the single task (walking) and the double task (walking and counting) using tailor-made software. Bigger difference between the parameters in both tasks indicates cognitive declines.

SECONDARY OUTCOMES:
Usability evaluation using video observations. | Day 1.
  Videos of the test procedure obtained from the target groups will be evaluated by usability experts.
  The video observations will be evaluated using the "Eisenhower's Urgent/Important Principle", in which items are evaluated as: "not urgent" - "urgent" and as "not important" - "important", whereby the "urgent" and the "important" items indicate higher needs of improvement.
Usability evaluation using questionnaire. | Day 1.
  Questionnaire addressing the personal experience with the screening procedure will be obtained from the target groups and will be evaluated by usability experts. The questionnaires will be evaluated using a score system (1-5), where 1 indicates very good usability.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Staubmann, MSc, Principal Investigator — FH Joanneum
Locations (1):
- FH-Joanneum, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Project homepage — https://scobes-ar.fh-joanneum.at
- See also: Eisenhower's Urgent/Important Principle: Using Time Effectively, Not Just Efficiently — http://www.mindtools.com